CLINICAL TRIAL: NCT00640003
Title: Baclofen Treatment of Ataxia Telangiectasia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NA_00002180
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Ataxia Telangiectasia
Keywords: AT; Ataxia; Telangiectasia
MeSH Terms: conditions — Ataxia Telangiectasia; Ataxia; Telangiectasis | interventions — Baclofen; Butyric Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Baclofen; Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: Baclofen; Drug: Placebo

INTERVENTIONS:
Drug: Baclofen — Drug given by orally via capsules. Escalation steps in 4-day intervals. Step 1: 5mg QAM. Step 2: 5mg BID. Step 3: 5mg TID. Step 4: 10mg QAM, 5mg BID. Step 5: 10mg BID, 5mg QMid-day. Step 6: 10mg TID. Step 6 will last up to 2 weeks. De-escalation will start from highest dose step and work backwards in 2-day intervals. Complete drug administration of escalating, staying constant at 10mg TID and de-escalating will be done with both drug and placebo.
  Other Names: Butanoic Acid
Drug: Placebo — placebo drug

SUMMARY:
This research is being done to find out if Baclofen, a medicine that is often used for the treatment of abnormal stiffness, might also be useful to treat some of the neurologic problems caused by ataxia telangiectasia (A-T). The investigators also want to find out if there are better ways to measure the problems of ataxia and abnormal eye movement for future studies of medication in ataxia telangiectasia.

ELIGIBILITY:
Inclusion Criteria:

* Teenagers over 12 years old and young adults with A-T may join if they have been evaluated previously in the A-T Clinical Center at Johns Hopkins Hospital and have a measurable abnormality of eye movement.
* Patients who are presently taking Baclofen will be eligible for the study if they are presently receiving the medication under the direction of Dr. Crawford in the ATCC, and are willing to withdraw from the medication for a period of one month prior to the initial screening visit.
* Female patients who are sexually active will be given a standard serum HCG pregnancy test.
* Those who are sexually active will be counseled about necessary precautions against pregnancy during the duration of the trial.

Exclusion Criteria:

* A positive pregnancy test.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Improvement in the decay constant for velocity storage as assessed by quantitative video examination of eye movement during and after rotation. | 3 months

SECONDARY OUTCOMES:
Other outcome measures include quantitative measurement of tremor, postural stability and a standard neurologic examination. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas O Crawford, M.D., Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States